CLINICAL TRIAL: NCT00554437
Title: Kenosha County Falls Prevention Study: An Intermediate-intensity, Community-based, Multifactorial Intervention
Brief Title: Kenosha County Falls Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Kenosha County Aging and Disability Resource Center (Other); Wisconsin Department of Health and Family Services (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-Prevention Funding
Record Dates: First submitted 2007-11-02; First posted 2007-11-06 (Estimated); Last update posted 2023-07-14 (Actual); Status verified 2008-11

CONDITIONS: Accidental Falls
Keywords: Accidental Falls; RCT; Age 65 and older; noninstitualized populations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intermediate-intensity, community-based, multifactorial falls intervention
  Interventions: Behavioral: UW Falls Prevention Program
- 2 (Active Comparator): Occupational therapist home safety evaluation
  Interventions: Behavioral: UW Falls Prevention Program

INTERVENTIONS:
Behavioral: UW Falls Prevention Program — The intervention model is of a community-based multifactorial intervention that links participants to existing medical care and service networks. The intervention used an algorithm based on the University of Wisconsin Falls Prevention Clinic, designed to identify predisposing factors for falls; induce risk reduction changes in medical conditions, medications, behavior, physical status, and home environment through recommendations to participants and their physicians; and make sure these changes are long-lasting through follow-up and linkages to other care networks.

SUMMARY:
Intensive falls prevention programs have been shown to be effective in reducing falls; however, a number of practical programs, based in community setting have not been successful at reducing rate of falls. The purpose of this study was to test, in a randomized, controlled trial, the efficacy of this intermediate-intensity, individual, multifactorial model to reduce falls. It was hypothesized that more contacts would lead to greater adherence and efficacy in reducing falls.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 and older
* a history of two falls in the previous year or one fall in the previous two years with injury or gait and balance problems
* independently living in Kenosha County

Exclusion Criteria:

* unable to give informed consent with no related caregiver in the home
* enrolled in hospice
* living in an assisted-living facility
* expecting to move away permanently from the area

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 349 (Actual)
Dates: Start 2002-05; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
rate of falls | one year

SECONDARY OUTCOMES:
all-cause hospitalizations | one year
nursing home utilizations: number of days and number of admissions | one year
change in ADL function from baseline to one year | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Mahoney, MD, Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- [Result] Mahoney JE, Shea TA, Przybelski R, Jaros L, Gangnon R, Cech S, Schwalbe A. Kenosha County falls prevention study: a randomized, controlled trial of an intermediate-intensity, community-based multifactorial falls intervention. J Am Geriatr Soc. 2007 Apr;55(4):489-98. doi: 10.1111/j.1532-5415.2007.01144.x. PMID 17397425